CLINICAL TRIAL: NCT02045602
Title: A Phase I, Multicenter, Open-label, Dose Escalation Study of Intravenous Administration of VCN-01 Oncolytic Adenovirus With or Without Gemcitabine and Abraxane® in Patients With Advanced Solid Tumors
Brief Title: Phase I Dose Escalation Study of Intravenous VCN-01 With or Without Gemcitabine and Abraxane® in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theriva Biologics SL (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-VCNA-001; 2012-005555-16 (EudraCT Number)
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors; Pancreatic Adenocarcinoma
Keywords: Cancer; Solid Tumors; Gemcitabine; Oncolytic virus; Metastatic; Pancreatic cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I: Dose Escalation, Single Agent (Experimental): Single intravenous injection of VCN-01 oncolytic adenovirus
  Interventions: Genetic: VCN-01
- Part II: Dose Escalation, Combination (Experimental): Single intravenous injection of VCN-01 oncolytic adenovirus in combination with Abraxane®/Gemcitabine
  Interventions: Genetic: VCN-01; Drug: Gemcitabine; Drug: Abraxane®
- Part III: Dose Escalation, Combination, "delayed" schedule (Experimental): Single intravenous injection of VCN-01 oncolytic adenovirus in combination with Abraxane®/Gemcitabine
  Interventions: Genetic: VCN-01; Drug: Gemcitabine; Drug: Abraxane®

INTERVENTIONS:
Genetic: VCN-01 — Genetically modified human adenovirus encoding human PH20 hyaluronidase
Drug: Gemcitabine — 1000 mg/m2 intravenous administration
  Arms: Part II: Dose Escalation, Combination; Part III: Dose Escalation, Combination, "delayed" schedule
Drug: Abraxane® — 125 mg/m2 intravenous administration
  Arms: Part II: Dose Escalation, Combination; Part III: Dose Escalation, Combination, "delayed" schedule

SUMMARY:
The purpose of this study is to determine the safety and tolerability of VCN-01 either administered alone or in combination with Abraxane®/Gemcitabine, and to determine the recommended phase II dose of VCN-01 alone or in combination with Abraxane®/Gemcitabine.

DETAILED DESCRIPTION:
The study consists of three parts:

* Part I is a dose escalation study to determine the safety and tolerability of a single intravenous injection of VCN-01 alone
* In Part II the safety and tolerability of the two highest VCN-01 tolerable doses from part I will be evaluated in combination with Abraxane®/Gemcitabine.
* In Part III the safety and tolerability of the two highest VCN-01 tolerable doses from part I will be evaluated in combination with Abraxane®/Gemcitabine in a "delayed" schedule compared with Part II.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female patients aged 18 years or over
* Patients must provide written informed consent
* Part I: Patients with histologically confirmed, locally advanced or metastatic solid tumors. Part II and Part III: Patients with histologically confirmed, pancreatic adenocarcinoma for which the established therapy is Abraxane®/Gemcitabine (clinical standard of care)
* Life expectancy above 3 months
* Patients willing to comply with treatment follow-up
* ECOG Performance status 0 or 1
* Adequate baseline organ function (hematologic, liver, renal and nutritional)
* Use a reliable method of contraception in fertile men and women

Exclusion Criteria:

* Active infection or other serious illness or autoimmune disease
* Treatment with live attenuated vaccines in the last three weeks
* Known chronic liver disease (liver cirrhosis, chronic hepatitis)
* Treatment with another investigational agent within its five half-lives prior to VCN-01 infusion
* Viral syndrome diagnosed during the two weeks before inclusion
* Chronic immunosuppressive therapy
* Concurrent malignant hematologic or solid disease
* Pregnancy or lactation. Patients must agree to use effective contraception or be surgically sterile.
* Patients receiving full-dose anticoagulant / antiplatelet therapy
* Adequate levels of neutralizing antibodies against adenovirus
* Patients with Li Fraumeni syndrome or with previous known retinoblastoma protein pathway germinal deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability by means of Adverse Events (AEs) and laboratory data | At least 6 months
Recommended Phase 2 Dose (RP2D) by determination of highest feasible dose (MFD) and any Dose Limiting Toxicities | At least 6 months

SECONDARY OUTCOMES:
Presence of VCN-01 in tumor | Day 8-10
  Determination of VCN-01 by analyzing viral genome copies in tumor biopsy
Viral Pharmacokinetics | Up to 48 h
  Determination of VCN-01 half-life by analyzing viral genome copies in blood
Viral Shedding | Up to day 28
  And at least up to 6 months follow-up in patients at the Maximum Tolerated Dose (MTD)
Neutralizing antibodies anti-VCN-01 | 30 days after end of treatment phase
  At least up to 6 months follow-up in patients at the MTD
Preliminary anti-tumor activity by Overall Response Rate (ORR) | CT or MRI scans every 8 weeks until disease progression
Preliminary anti-tumor activity by Progression Free Survival (PFS) | CT or MRI scans every 8 weeks until disease progression

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Derived] Garcia-Carbonero R, Bazan-Peregrino M, Gil-Martin M, Alvarez R, Macarulla T, Riesco-Martinez MC, Verdaguer H, Guillen-Ponce C, Farrera-Sal M, Moreno R, Mato-Berciano A, Maliandi MV, Torres-Manjon S, Costa M, Del Pozo N, Martinez de Villarreal J, Real FX, Vidal N, Capella G, Alemany R, Blasi E, Blasco C, Cascallo M, Salazar R. Phase I, multicenter, open-label study of intravenous VCN-01 oncolytic adenovirus with or without nab-paclitaxel plus gemcitabine in patients with advanced solid tumors. J Immunother Cancer. 2022 Mar;10(3):e003255. doi: 10.1136/jitc-2021-003255. PMID 35338084